CLINICAL TRIAL: NCT00640029
Title: Medico-economic Evaluation of the Prosthetic Replacement of the Lumbar and Cervical Intervertebral Disc
Brief Title: Evaluation of the Prosthetic Disc Replacement
Acronym: EVA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insuffisent recruitment
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P060409
Record Dates: First submitted 2008-02-15; First posted 2008-03-20 (Estimated); Last update posted 2015-03-10 (Estimated); Status verified 2015-03

CONDITIONS: Lumbar Degenerative Disc Disease; Cervical Degenerative Disc Disease; Kyphosis
Keywords: Arthroplasty; Arthrodesis; Prosthesis; Disc replacement; Spine; Lumbar; Cervical; Intervertebral disk; Cervical or lumbar intervertebral disk; Degenerative pathology
MeSH Terms: conditions — Intervertebral Disc Degeneration; Kyphosis; Ankylosis | interventions — Arthrodesis; Arthroplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- 1 (Experimental): Cervical - Arthroplasty
  Interventions: Device: Arthroplasty (PRODISC-C® , PRODISC-L®, Mobi-C®, Mobidisc®, PrestigeLP®, A-Mav®, O-Mav®, DISCOCERV®)
- 2 (Active Comparator): Cervical - Arthrodesis
  Interventions: Procedure: Arthrodesis
- 3 (Experimental): Lumbar - Over 50 years - Arthroplasty
  Interventions: Device: Arthroplasty (PRODISC-C® , PRODISC-L®, Mobi-C®, Mobidisc®, PrestigeLP®, A-Mav®, O-Mav®, DISCOCERV®)
- 4 (Active Comparator): Lumbar - Over 50 years - Arthrodesis
  Interventions: Procedure: Arthrodesis
- 5 (Experimental): Lumbar - Under 50 years - Arthroplasty
  Interventions: Device: Arthroplasty (PRODISC-C® , PRODISC-L®, Mobi-C®, Mobidisc®, PrestigeLP®, A-Mav®, O-Mav®, DISCOCERV®)

INTERVENTIONS:
Procedure: Arthrodesis — * posterior,
  * anterior,
  * circumference approach
  Arms: 2; 4
Device: Arthroplasty (PRODISC-C® , PRODISC-L®, Mobi-C®, Mobidisc®, PrestigeLP®, A-Mav®, O-Mav®, DISCOCERV®) — * SYNTHES : PRODISC-C® , PRODISC-L®
  * LDR : Mobi-C®, Mobidisc®
  * MEDTRONIC : PrestigeLP®, A-Mav®, O-Mav®
  * SCIENT'X : DISCOCERV®
  Arms: 1; 3; 5

SUMMARY:
Until now, arthrodesis (intervertebral fusion) is the formal treatment for the lumbar and cervical degenerative disc disease : arthrodesis has been the standard surgical treatment for the patients when nonsurgical management has failed. However , it has shown out some drawbacks : pseudoarthrosis may appear in the short term, and junctional degeneration in the long term.

The replacement of the intervertebral disc by a prosthesis (arthroplasty) has been since a few years a major alternative therapeutic to the arthrodesis.: it demonstrates great functional results and less post-interventional complications. It is indicated to restore a normal function of the spine (motion is kept)and to avoid deterioration of the adjacent spinal segments over the long time.

In this clinical study, we will distinguish the cervical discal pathology and the lumbar discal pathology.

The purpose of this study is to analyze the results of the arthroplasty in terms of functional effects, quality of life, anatomical results and economical results.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the cervical and lumbar intervertebral disc replacement by a prosthesis ( arthroplasty ) in adults suffering from degenerative disc disease.

For the cervical pathology, a comparative randomized multi-site study of the medico-economic evaluation of the prosthesis implementation versus arthrodesis, the standard treatment, will be realised , for patients from 20 to 55 years old, within very rigorous exclusion and inclusion criteria.

For the lumbar pathology, a comparative randomized multi-site study of the medico-economic evaluation of the prosthesis implementation versus arthrodesis, the standard treatment, will be realized , for patients from 50 to 65 years old, within acute exclusion and inclusion criteria.

For patients under 50 years old, randomization is not used as arthroplasty offers very good results. By these young patients, a cohort study will thus be realized.

Patients with degenerative discal disease at one or more levels will be recruited in 17 sites in France :

* 3 sites in ASSITANCE PUBLIQUE - HOPITAUX DE PARIS (AP-HP)
* 14 sites in France outside AP-HP.

The study will have 3 parts :

* Cervical pathology : 500 patients divided on 250 arthroplasties and 250 arthrodeses.
* Lumbar pathology : 525 patients divided according to their age:
* over 50 years old : randomization in 175 lumbar arthroplasties and 175 lumbar arthrodeses.
* until 50 years old : cohort study : 175 lumbar arthroplasties.

This study will last 3 years : a 2 year-period of inclusion , and a post interventional one year-follow-up period for each included patient.

The duration of the participation in the study for each patient is one year.

7 evaluations will be realized for each patient : pre-interventional visit, intervention, post-interventional visit, visit at 45 days, visit at 3 months, visit at 6 months and visit at one year.

Each visit will comprise different exams and observations.

The criterion of principle judgement will be the quality of life measured as follows :

* For the lumbar pathology, the Oswestry Low Back Pain Disability Questionnaire, the SF36 Questionnaire, the Visual Analog Scale (Pain), at each visit.
* For the cervical pathology : the NDI score, the SF36 Questionnaire, the Visual Analog Scale (Pain), at each visit.

The secondary criteria will be medico-economical and clinical too. Arthrodesis and Arthroplasty will be compared in terms of:

* anatomical results of the intervention
* intervention tolerance
* wear (estimated by the discal height)
* costs of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* cervical disc:

  * 20 to 55 years old;
  * symptomatic disc disease between C3-C7 defined as:
  * Cervical or brachial(radicular) pain and/or functional/neurologic deficit with at least one of the following conditions confirmed by imaging :
  * Hernia of the gelatinous core;
  * Spondylosis (osteophytes); loss of height of the disc;
  * Not reacting to the no-invasive treatment or progressive symptoms or compressions ;
  * NDI >= 15/50;
  * Ready to respect the instructions;
  * More than one vertebral level requiring a treatment;
  * At a vertebral block close to the level to be treated;
  * Associated to a fusion at the adjacent level or another level;
  * Written assent;
  * Patient who can receive one or other treatment;
* lumbar disc:

  * 25 to 65 years;
  * Symptomatology of prevalent lumbago with or without radiculalgia and failure of the medical treatments;
  * Idiopathic discopathies or after cure of disc herniations (except prior infections);
  * Repetition of disc herniation (except excluded hernia);
  * Discopathies with median posterior disc herniation with limited development and loss of discal height;
  * 1 or 2 contiguous stages or not among L3L4, L4L5, L5S1;
  * Written assent;
  * Patient who can receive one or other treatment;

Exclusion Criteria:

* cervical disc:

  * Cervical instability: in flexion/extension Translation > 3 mm and /or >11 degrees of rotary difference with one or the other adjacent level;
  * Serious problem of articular facet or degeneration.;
  * Known allergy to cobalt, chromium plates, molybdenum, titanium or polyethylene;
  * Clinically compromised vertebrae at level (s) touched after a current or passed traumatism;
  * Serious spondylosis (MESOCEPHALES osteophytes; loss height of the disc>70% or Absence of motion(< 2°));
  * Osteoporosis(DEXA);
  * Paget, osteomalacia or metabolic osseous disturbs ;
  * Serious Willis disease asking an insulin management;
  * Pregnancy;
  * Active, local or generalized infection;
  * Taking treatments or drugs which one knows that they interfere on the management of the bone/ the soft part (e.g. steroids);
  * Rheumatoid arthritis or another disease car-immune;
  * Systemic disease (AIDS, HIV, hepatitis);
  * Active malignity compromising the vital forecast at the short term;
  * Septic antecedents;
  * No-affiliation with the Social Security;
  * Patient refusing to be recontacted by mail or telephone apart from the visits;
  * Patient refusing the randomization;
* lumbar disc:

  * Morbid Obesity;
  * Abdomen multi operated;
  * Crowned slope L5-S1 high;
  * Traumatic after-effects with moderate deformations of the vertebra ;
  * Symptomatic lumbar canal stenosis;
  * Septic antecedents of the site to be operated;
  * Great degenerative or constitutional vertebral instability ;
  * Narrow lumbar channel and/or excluded and migrated lumbar slipped disc;
  * Scoliosis >8;
  * Advanced articular osteoarthritis;
  * Severe osteoporosis ;
  * Disease of Paget, Osteomalacia, disturb metabolic osseous;
  * Disease car-immune rheumatoid;
  * Pregnancy;
  * Badly balanced diabetes ;
  * Systemic disease;
  * Vascular Problem (arteritis lower limb, aortic aneurism);
  * Evolutionary Hepatitis ;
  * Immunodeficient Disease (of which HIV);
  * No-affiliation with the Social Security;
  * Patient refusing to be recontacted by mail or telephone apart from the visits;
  * Patient refusing the randomization;

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 301 (Actual)
Dates: Start 2008-02; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction at one year. Oswestry questionnaire (lumbar pathology) or NDI questionnaire (cervical pathology), SF36 score and Visual Analog Scale (Pain | 1 year

SECONDARY OUTCOMES:
Patient satisfaction at post-interventional visit, after 45 days, at 3 months, and at 6 months | post-interventional visit, after 45 days, at 3 months, at 6 months and 1 year
Cost of the treatments | post-interventional visit, after 45 days, at 3 months, at 6 months and 1 year
Tolerance of the intervention, stability of the prosthesis | post-interventional visit, after 45 days, at 3 months, at 6 months and 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Cottin, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Jacques BRUNON, MD, PhD, Principal Investigator — Saint-Etienne's Hospital
Locations (2):
- France (2):
  - Service de Chirurgie CHU Hopital Antoine Béclère, Clamart
  - Service de Neurochirurgie CHU Saint-Etienne, Saint-Etienne